CLINICAL TRIAL: NCT04936815
Title: Effectiveness of Echocardiographic Screening of Pregnant Women During Antenatal Care
Brief Title: Echocardiographic Screening of Pregnant Women During Antenatal Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Pilgrim (Other)
Collaborators: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Thomas Pilgrim, Deputy Physician-in-Chief, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRC/2121/021
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Valvular Heart Disease; Rheumatic Heart Disease; Pregnancy Complications
MeSH Terms: conditions — Heart Valve Diseases; Rheumatic Heart Disease; Pregnancy Complications | interventions — Echocardiography

STUDY DESIGN:
Intervention Model Description: Three clusters representing the three administrative units of the Ob/Gyn department will be randomly allocated to an experimental or a control condition. During 18 months, each of the three clusters will undergo a randomly allocated experimental period of 6 months and two control periods of 6 months. Women seen at least once during the experimental period will be offered to undergo systematic echocardiographic screening for structural heart disease followed by guideline-directed peripartum management. Women only seen during the control periods will undergo routine antenatal care and receive echocardiography only if clinically indicated. After 15 months recruitment, the investigators will perform a conditional power analysis. If the conditional power is below 80% but above 50%, and an extension is considered feasible, the investigators will extend the recruitment duration to 36 months and allocate each administrative unit to another experimental recruitment period of 6 months duration.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echocardiographic screening (Experimental): Echocardiographic screening for the detection of latent structural heart disease
  Interventions: Diagnostic Test: Transthoracic echocardiography
- Control arm (No Intervention): Routine antenatal care

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Transthoracic echocardiography for the detection of congenital or acquired structural heart disease.
  Arms: Echocardiographic screening

SUMMARY:
Non-obstetrical drivers of adverse pregnancy outcomes are underappreciated. Latent structural heart disease may account for a substantial proportion of adverse pregnancy outcomes in low-resource settings.

Pregnant women presenting to B.P. Koirala Institute of Health Sciences will be prospectively included into a registry upon their visit for antenatal care. Women will be followed until 6 weeks after the time of delivery. Nested within this registry, the investigators will perform a registry-based adaptive cluster randomized crossover trial. The trial compares an experimental condition (echocardiographic screening) and a control condition (routine antenatal care).

DETAILED DESCRIPTION:
Latent structural heart disease may result in complications during pregnancy and delivery. Echocardiographic screening of pregnant women allows for timely detection of structural heart disease in women that may complicate delivery and jeopardize the health and well-being of both the mother and the newborn. In a setting of high rates of latent rheumatic heart disease, with particular high prevalence among women, systematic echocardiographic screening may be a pragmatic approach to prevent adverse clinical outcome related to valvular heart failure. Systematic echocardiographic screening proved to be effective among children in endemic regions.

The present study is a registry-based, adaptive cluster randomized crossover trial. The trial will be nested into a registry of pregnant women presenting for routine antenatal care. The experimental condition will be echocardiographic screening. The control condition will be no echocardiographic screening.

In the experimental condition, all pregnant women presenting for routine antenatal care will be offered transthoracic echocardiographic screening for the detection of latent structural heart disease. In the control condition, pregnant women will undergo routine antenatal care with echocardiography only when clinically indicated. Ascertainment of the primary endpoint will be performed at hospital discharge after delivery and will rely on routinely collected data. All events will be independently adjudicated by an expert panel of pediatricians, cardiologists and gynecologists.

The randomization relates solely to the detection of rheumatic heart disease, while treatment follows guideline recommendations. It is important to note, that all women both in the experimental arm and the control arm detected to have heart disease will undergo optimal medical management during pregnancy and delivery according to the most recent guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥18 years presenting for routine antenatal care.
* Written informed consent.

Exclusion Criteria:

* Women presenting to the hospital after delivery.
* Women presenting directly for delivery without previous antenatal care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint | For APGAR Score: 10 minutes after birth. For all other components of the composite endpoint: Hospital discharge after delivery (on an average of 4 days after delivery) or 7 days after delivery (whatever takes first).
  Incidence rate of the composite of maternal death, fetal/neonatal death, maternal heart failure, maternal hospitalization for cardiovascular reasons or an APGAR Score <7.

SECONDARY OUTCOMES:
Incidence of maternal adverse events | 6 weeks after delivery
  Death; Cerebrovascular Events; Heart failure; Cardiac interventions; Supraventricular tachycardia, Atrial fibrillation, Ventricular tachycardia; Thrombotic and thromboembolic events; Postpartum haemorrhage.
Incidence of fetal/neonatal adverse events | 6 weeks after delivery
  Death; Preterm birth (<37 weeks); Birthweight <2500g

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, MSc, Principal Investigator — Department of Cardiology, Bern University Hospital, Switzerland
Locations (2):
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No